CLINICAL TRIAL: NCT04890028
Title: Detection and Metabolic Characterization in DOPA PET/CT of no Treated Brain Metastases of Lung Cancer, Breast Cancer and Melanoma
Brief Title: Detection and Metabolic Characterization in DOPA PET/CT of Brain Metastases
Acronym: DOPACER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Cancerologie de l'Ouest (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ICO-2020-28
Record Dates: First submitted 2021-05-12; First posted 2021-05-18 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-07

CONDITIONS: Brain Metastases; MRI
Keywords: Breast cancer; Lung Cancer; Melanoma; DOPA PET/CT
MeSH Terms: conditions — Brain Neoplasms; Breast Neoplasms; Lung Neoplasms; Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- F-DOPA PET/CT (Experimental): Drug: 18 F-DOPA Radiation: F-DOPA PET CT
  Interventions: Radiation: F-DOPA PET/CT

INTERVENTIONS:
Radiation: F-DOPA PET/CT — All subjects will be imaged
  1 time injection of 2 MBq/kg of 18F-DOPA

SUMMARY:
About 20 to 30% of patients treated for cancer will have brain metastases. These brain metastases are found more frequently in patients with lung cancer, breast cancer or melanoma. The prognosis of these patients is unfavorable but prolonged survival can be obtained with the local and systemic treatments currently available.

Brain MRI is the gold standard for evaluating brain metastases but has limitations in therapeutic evaluation, partially offset by PET imaging of amino acid metabolism.

Our work aims to compare the performance of PET-DOPA with standard MRI for the detection of brain metastases (≥ 5mm) in lung cancer, breast cancer and melanoma; and to characterize these lesions using dynamic acquisitions obtained with a digital PET camera with high spatial resolution. Having better knowledge of the metabolic characteristics of newly discovered brain metastases, the objective of subsequent studies will be to better assess the per- or post-therapeutic efficacy of radiotherapy and the various systemic therapies available (chemotherapy, targeted therapy, immunotherapy).

ELIGIBILITY:
Inclusion Criteria:

* Primitive cancer (brest cancer, lung cancer, melanoma) proven histologically
* Presence of brain metastasis visualized on MRI, of which at least one measures 5 mm
* Age > 18 years
* Patient has valid health insurance
* Written informed consent obtained from the patient prior to performing any protocol-related procedures, including screening evaluations

Exclusion Criteria:

* History of irradiation cerebral
* History of brain surgery for brain metastasis or glial tumor
* Systemic therapy (chemotherapy, targeted therapy, immunotherapy) modified in the 6 weeks preceding the realization of DOPA PET/CT,
* New anti-tumor treatment started between the discovery of brain metastases and the performance of DOPA PET/CT
* Other concomitant cancer, or history of cancer in the 5 years preceding the performance of DOPA PET/CT
* Pregnant or lactating females
* Persons deprived of their liberty, under a measure of safeguard of justice, under guardianship or placed under the authority of a guardian.

Disorder precluding understanding of trial information or informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2021-12-03 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Assess the sensitivity of 18F DOPA PET-CT for the detection of no treated brain metastases (breast cancer, lung cancer, melanoma), newly diagnosed by MRI and measuring at least 5 mm in diameter. | Within 8 months of PET-CT
  The sensitivity of PET-DOPA to detect brain metastases greater than 5 mm is determined by the number of metastases detected with PET-DOPA compared to the number of metastases greater than 5 mm detected by MRI

SECONDARY OUTCOMES:
Assess the sensitivity of 18F DOPA PET-CT according to the site of the primary tumor (lung cancer, breast cancer, melanoma) and its characteristics | Within 8 months of PET-CT
  The sensitivity per site will be calculated for 8 primary tumor categories: 3 for lung cancer (EGFR mutation or ALK rearrangement; PDL1 +; others), 2 for melanoma (BRAF V600 mutation; others), 3 for breast cancer (triple negative; Her2 + RH-; others)

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Morel, MD, Principal Investigator — Institut de Cancérologie de l'Ouest
Locations (3):
- France (3):
  - CHU Angers, Angers
  - Institut de Cancerologie de l'Ouest, Angers
  - Institut de Cancerologie de L'Ouest, Saint-Herblain

IPD SHARING:
Plan to Share IPD: No